CLINICAL TRIAL: NCT03018028
Title: Dose-response, Safety and Efficacy of Oral Semaglutide Versus Placebo and Versus Liraglutide, All as Monotherapy in Japanese Subjects With Type 2 Diabetes
Acronym: PIONEER 9
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9924-4281; U1111-1181-4048 (Other: WHO); JapicCTI-173489 (Other: JAPIC)
Record Dates: First submitted 2017-01-06; First posted 2017-01-11 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Oral semaglutide 3 mg (Experimental)
  Interventions: Drug: Semaglutide
- Oral semaglutide 7 mg (Experimental)
  Interventions: Drug: Semaglutide
- Oral semaglutide 14 mg (Experimental)
  Interventions: Drug: Semaglutide
- Oral placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Liraglutide 0.9 mg (Active Comparator)
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Semaglutide — Oral administration once daily
  Arms: Oral semaglutide 14 mg; Oral semaglutide 3 mg; Oral semaglutide 7 mg
Drug: Placebo — Oral administration once daily
  Arms: Oral placebo
Drug: Liraglutide — Subcutaneous (s.c., under the skin) injection once daily
  Arms: Liraglutide 0.9 mg

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to investigate the dose-response relationship of once-daily dosing of three dose levels (3, 7 and 14 mg) of oral semaglutide versus placebo as monotherapy on glycaemic control in Japanese subjects with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Japanese male or female, age above or equal to 20 years at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus for at least 30 days prior to day of screening
* HbA1c 6.5%-9.5% (48-80 mmol/mol) (both inclusive) for subjects treated with oral antidiabetic drug as monotherapy and 7.0%-10.0% (53-86 mmol/mol) (both inclusive) for subjects treated with diet and exercise therapy alone
* Treatment for at least 30 days prior to day of screening with;- stable daily dose of oral anti-diabetic drug as monotherapy (allowed oral anti-diabetic drugs are: metformin, sulphonylurea, glinide, α-glucosidase inhibitor, dipeptidyl peptidase-4 inhibitor and sodium-glucose cotransporter-2 inhibitor) at a half-maximum approved dose or below according to Japanese labelling in addition to diet and exercise therapy. or - diet and exercise therapy alone

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method. Adequate contraceptive measures are abstinence (not having sex), diaphragm, condom (by the partner), intrauterine device, sponge, spermicide or oral contraceptives
* Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol
* Family or personal history of multiple endocrine neoplasia type 2 (MEN 2) or medullary thyroid carcinoma (MTC)
* History of pancreatitis (acute or chronic)
* History of major surgical procedures involving the stomach and potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery)
* Any of the following: myocardial infarction, stroke or hospitalisation for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening and randomisation
* Subject presently classified as being in New York Heart Association (NYHA) Class IV
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* Subjects with alanine aminotransferase (ALT) above 2.5 x upper normal limit (UNL)
* Renal impairment defined as estimated Glomerular Filtration Rate (eGFR) below 30 mL/min/1.73 m^2 as per Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI)
* Treatment with once-weekly glucagon-like peptide-1 receptor agonist (GLP-1 RA), once weekly dipeptidyl peptidase-4 (DPP-4) inhibitor or thiazolidinedione in a period of 90 days before the day of screening
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 60 days before the day of screening. An exception is short-term insulin treatment for acute illness for a total of below or equal to 14 days
* Proliferative retinopathy or maculopathy requiring acute treatment. Verified by fundus photography or dilated fundoscopy performed within 90 days prior to randomisation
* History or presence of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer and in-situ carcinomas)
* Initiation of anti-diabetic medication between the day of screening and the day of randomisation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Japan (13):
  - Novo Nordisk Investigational Site, Akita-shi, Akita
  - Novo Nordisk Investigational Site, Arakawa-ku, Tokyo
  - Novo Nordisk Investigational Site, Ebina-shi, Kanagawa
  - Novo Nordisk Investigational Site, Gunma
  - Novo Nordisk Investigational Site, Kanagawa
  - Novo Nordisk Investigational Site, Minato-ku, Tokyo
  - Novo Nordisk Investigational Site, Naka
  - Novo Nordisk Investigational Site, Osaka-shi, Osaka
  - Novo Nordisk Investigational Site, Ota-ku, Tokyo
  - Novo Nordisk Investigational Site, Saga-shi, Saga
  - Novo Nordisk Investigational Site, Sendai-shi, Miyagi
  - Novo Nordisk Investigational Site, Suita-shi, Osaka
  - Novo Nordisk Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Derived] Husain M, Bain SC, Holst AG, Mark T, Rasmussen S, Lingvay I. Effects of semaglutide on risk of cardiovascular events across a continuum of cardiovascular risk: combined post hoc analysis of the SUSTAIN and PIONEER trials. Cardiovasc Diabetol. 2020 Sep 30;19(1):156. doi: 10.1186/s12933-020-01106-4. PMID 32998732
- [Derived] Yamada Y, Katagiri H, Hamamoto Y, Deenadayalan S, Navarria A, Nishijima K, Seino Y; PIONEER 9 investigators. Dose-response, efficacy, and safety of oral semaglutide monotherapy in Japanese patients with type 2 diabetes (PIONEER 9): a 52-week, phase 2/3a, randomised, controlled trial. Lancet Diabetes Endocrinol. 2020 May;8(5):377-391. doi: 10.1016/S2213-8587(20)30075-9. PMID 32333875
- [Derived] Thethi TK, Pratley R, Meier JJ. Efficacy, safety and cardiovascular outcomes of once-daily oral semaglutide in patients with type 2 diabetes: The PIONEER programme. Diabetes Obes Metab. 2020 Aug;22(8):1263-1277. doi: 10.1111/dom.14054. Epub 2020 May 13. PMID 32267058
- [Derived] Husain M, Bain SC, Jeppesen OK, Lingvay I, Sorrig R, Treppendahl MB, Vilsboll T. Semaglutide (SUSTAIN and PIONEER) reduces cardiovascular events in type 2 diabetes across varying cardiovascular risk. Diabetes Obes Metab. 2020 Mar;22(3):442-451. doi: 10.1111/dom.13955. Epub 2020 Feb 5. PMID 31903692

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 16 sites in Japan. Japanese participants with type 2 diabetes (T2D) treated with either diet and exercise alone or with oral anti-diabetic drug (OAD) monotherapy for at least 30 days prior to screening were enrolled in the study.
Pre-assignment Details: Data presented in "participant flow" is based on the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Groups:
- Oral Semaglutide 3 mg: Participants received 3.0 milligrams (mg) of oral semaglutide tablets once daily in the morning in fasted state for 52 weeks. The oral semaglutide tablet was taken once daily in a fasting state at least 30 min before the first meal of the day with up to half a glass of water.
- Oral Semaglutide 7 mg: Participants received oral semaglutide tablets once daily in the morning in fasted state for 52 weeks. Participants started oral semaglutide at 3 mg and were dose escalated in 4-week increments until the final maintenance dose of 7 mg once-daily was reached (i.e. 3 mg from week 0 to week 4, 7 mg from week 4 to week 52). The oral semaglutide tablet was taken once daily in a fasting state at least 30 min before the first meal of the day with up to half a glass of water.
- Oral Semaglutide 14 mg: Participants received oral semaglutide tablets once daily in the morning in fasted state for 52 weeks. Participants started oral semaglutide at 3 mg and were dose escalated in 4-week increments until the final maintenance dose of 14 mg once-daily was reached (i.e. 3 mg from week 0 to week 4, 7 mg from week 4 to week 8, 14 mg from week 8 to week 52). The oral semaglutide tablet was taken once daily in a fasting state at least 30 min before the first meal of the day with up to half a glass of water.
- Liraglutide 0.9 mg: Participants received liraglutide for 52 weeks. Liraglutide was administered once-daily as subcutaneous injection (under the skin) in the abdomen, thigh or upper arm and was taken with or without food, preferably at the same time in the morning or evening. Participants initiated liraglutide at 0.3 mg once-daily, and were dose escalated after 1 week to 0.6 mg, and then dose escalated after 1 week to the recommended maximum dose of 0.9 mg.
- Placebo: Participants received placebo (for oral semaglutide) tablets once daily for 52 weeks. The placebo tablet was taken once daily in the morning in a fasting state at least 30 min before the first meal of the day with up to half a glass of water.
Period: Overall Study
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Started | 49 | 49 | 48 | 48 | 49
Full Analysis Set (FAS) | 49 | 49 | 48 | 48 | 49
Safety Analysis Set (SAS) | 49 | 49 | 48 | 48 | 49
Completed | 46 | 49 | 47 | 46 | 49
Not Completed | 3 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on full analysis set, which included all randomised participants.
Groups:
- Oral Semaglutide 3 mg: Participants received 3.0 mg of oral semaglutide tablets once daily in the morning in fasted state for 52 weeks. The oral semaglutide tablet was taken once daily in a fasting state at least 30 min before the first meal of the day with up to half a glass of water.
- Total: Total of all reporting groups
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo | Total
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49 | 243
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58 (9) | 60 (10) | 61 (9) | 59 (10) | 59 (9) | 59 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 8 | 9 | 9 | 52
  Male | 36 | 36 | 40 | 39 | 40 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 49 | 49 | 48 | 48 | 49 | 243
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 49 | 49 | 48 | 48 | 49 | 243
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Baseline HbA1c [Mean (Standard Deviation); unit: Percentage of HbA1c] — Observed mean HbA1c
  Percentage of HbA1c | 8.1 (0.8) | 8.3 (1.0) | 8.0 (0.9) | 8.3 (0.8) | 8.3 (1.1) | 8.2 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Week 26)
Description: Change from baseline (week 0) to week 26 in glycosylated haemoglobin (HbA1c). The endpoint was analysed based on data from the on-treatment without rescue medication observation period. On-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication. The endpoint was also evaluated based on data from the in-trial observation period. In-trial observation period - time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = full analysis set (FAS) which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Percentage point of HbA1c
  On-treatment without rescue medication: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  On-treatment without rescue medication | -1.1 (0.8) | -1.7 (0.8) | -1.7 (0.8) | -1.4 (1.1) | -0.2 (0.7)
  In-trial observation period: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  In-trial observation period | -1.1 (0.8) | -1.6 (0.8) | -1.7 (0.9) | -1.4 (1.1) | -0.4 (1.0)
Statistical Analysis 1: Comparison: Oral Semaglutide 3 mg vs Placebo; The analysis was based on a mixed model for repeated measurements (MMRM) that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment and stratification factor as categorical fixed effects and the baseline HbA1c value as a covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Superiority — This hypothesis was not controlled for multiplicity. Results are based on the data from the on-treatment without rescue medication observation period. The estimated treatment effect excludes the effect of any rescue medication and any effect after premature trial product discontinuation (hypothetical estimand); p < 0.0001, Mixed model for repeated measurements — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -1.1, 95% CI 2-sided [-1.4 to -0.8] — Oral semaglutide 3 mg - Placebo
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Placebo; The analysis was based on a MMRM that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment and stratification factor as categorical fixed effects and the baseline HbA1c value as a covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed model for repeated measurements — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -1.5, 95% CI 2-sided [-1.7 to -1.2] — Oral semaglutide 7 mg - Placebo
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed model for repeated measurements — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -1.7, 95% CI 2-sided [-2.0 to -1.4] — Oral semaglutide 14 mg - Placebo
Statistical Analysis 4: Comparison: Oral Semaglutide 3 mg vs Liraglutide 0.9 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0799, Mixed model for repeated measurements — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = 0.3, 95% CI 2-sided [-0.0 to 0.6] — Oral semaglutide 3 mg - Liraglutide 0.9 mg
Statistical Analysis 5: Comparison: Oral Semaglutide 7 mg vs Liraglutide 0.9 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3942, Mixed model for repeated measurements — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -0.1, 95% CI 2-sided [-0.4 to 0.2] — Oral semaglutide 7 mg - Liraglutide 0.9 mg
Statistical Analysis 6: Comparison: Oral Semaglutide 14 mg vs Liraglutide 0.9 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0272, Mixed model for repeated measurement — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -0.3, 95% CI 2-sided [-0.6 to -0.0] — Oral semaglutide 14 mg - Liraglutide 0.9 mg
Statistical Analysis 7: Comparison: Oral Semaglutide 3 mg vs Placebo; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 26 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using an analysis of covariance (ANCOVA) model with treatment and stratification factor as categorical fixed effects and baseline HbA1c as a covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Superiority — This hypothesis was not controlled for multiplicity. Results are based on the data from the in-trial observation period. The estimated treatment effect includes the effect of any rescue medication and any effect after premature trial product discontinuation (treatment policy estimand); p < 0.0001, Pattern Mixture model — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -0.8, 95% CI 2-sided [-1.1 to -0.5] — Oral semaglutide 3 mg - Placebo
Statistical Analysis 8: Comparison: Oral Semaglutide 7 mg vs Placebo; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 26 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using an ANCOVA model with treatment and stratification factor as categorical fixed effects and baseline HbA1c as a covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Superiority — [test comment as in outcome 1, analysis 7]; p < 0.0001, Pattern Mixture model — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -1.2, 95% CI 2-sided [-1.5 to -0.9] — Oral semaglutide 7 mg - Placebo
Statistical Analysis 9: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 1, analysis 8]; Test type: Superiority — [test comment as in outcome 1, analysis 7]; p < 0.0001, Pattern Mixture model — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -1.4, 95% CI 2-sided [-1.7 to -1.1] — Oral semaglutide 14 mg - Placebo
Statistical Analysis 10: Comparison: Oral Semaglutide 3 mg vs Liraglutide 0.9 mg; [analysis description as in outcome 1, analysis 8]; Test type: Superiority — [test comment as in outcome 1, analysis 7]; p = 0.1958, Pattern Mixture model — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = 0.2, 95% CI 2-sided [-0.1 to 0.5] — Oral semaglutide 3 mg - Liraglutide 0.9 mg
Statistical Analysis 11: Comparison: Oral Semaglutide 7 mg vs Liraglutide 0.9 mg; [analysis description as in outcome 1, analysis 8]; Test type: Superiority — [test comment as in outcome 1, analysis 7]; p = 0.1868, Pattern Mixture model — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -0.2, 95% CI 2-sided [-0.5 to 0.1] — Oral semaglutide 7 mg - Liraglutide 0.9 mg
Statistical Analysis 12: Comparison: Oral Semaglutide 14 mg vs Liraglutide 0.9 mg; [analysis description as in outcome 1, analysis 8]; Test type: Superiority — [test comment as in outcome 1, analysis 7]; p = 0.0077, Pattern Mixture model — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -0.4, 95% CI 2-sided [-0.7 to -0.1] — Oral semaglutide 14 mg - Liraglutide 0.9 mg

2. Secondary Outcome: Change in HbA1c (Week 52)
Description: Change from baseline (week 0) to week 52 in HbA1c. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
Percentage of HbA1c | -1.0 (0.9) | -1.4 (0.9) | -1.5 (0.8) | -1.3 (1.0) | 0.1 (0.7)

3. Secondary Outcome: Change in Body Weight (kg)
Description: Change from baseline (week 0) in body weight. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: Overall number of participants analyzed = FAS which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Kilogram (kg)
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26 | -0.4 (1.9) | -1.2 (1.9) | -2.4 (3.0) | 0.1 (1.6) | -1.1 (1.6)
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52 | 0.0 (2.4) | -0.8 (2.1) | -2.9 (3.9) | 0.5 (2.0) | -1.0 (1.7)

4. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change from baseline (week 0) in fasting plasma glucose. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Millimoles per liter (mmol/L)
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26 | -1.62 (1.74) | -1.60 (1.74) | -2.37 (1.84) | -2.48 (1.76) | -0.37 (1.50)
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52 | -1.13 (1.82) | -1.60 (1.22) | -2.29 (1.62) | -2.28 (2.09) | 0.33 (1.31)

5. Secondary Outcome: Change in Self-measured Plasma Glucose 7-point Profile (SMPG) - Mean 7-point Profile
Description: Change from baseline (week 0) in mean 7-point self-measured plasma glucose (SMPG) profile. SMPG was recorded at the following 7 time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after dinner and at bedtime. Mean 7-point profile was defined as the area under the profile, calculated using the trapezoidal method, divided by the measurement time. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
mmol/L
  Week 26: number analyzed (Participants) | 43 | 46 | 44 | 44 | 42
  Week 26 | -2.2 (2.2) | -2.6 (1.8) | -3.1 (2.1) | -2.8 (2.1) | -0.8 (1.7)
  Week 52: number analyzed (Participants) | 37 | 43 | 41 | 39 | 34
  Week 52 | -1.7 (1.7) | -2.2 (1.9) | -3.1 (2.1) | -2.3 (2.5) | -0.0 (1.7)

6. Secondary Outcome: Change in Mean Postprandial Increment Over All Meals in SMPG
Description: Change from baseline (week 0) in the average of the post-prandial increments over all meals. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
mmol/L
  Week 26: number analyzed (Participants) | 43 | 46 | 44 | 44 | 42
  Week 26 | -0.7 (2.1) | -1.2 (2.3) | -2.0 (2.3) | -1.1 (2.1) | -0.5 (2.4)
  Week 52: number analyzed (Participants) | 37 | 43 | 41 | 39 | 34
  Week 52 | -0.5 (2.4) | -0.9 (2.4) | -2.0 (2.1) | -0.6 (2.2) | -0.1 (2.4)

7. Secondary Outcome: Change in Body Weight (%)
Description: Relative change (%) from baseline (week 0) in body weight (kg). Data based on on-treatment without resue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Percentage change
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26 | -0.64 (2.65) | -1.63 (2.78) | -3.54 (4.33) | 0.08 (2.23) | -1.58 (2.27)
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52 | -0.03 (3.25) | -1.23 (3.09) | -4.42 (5.91) | 0.68 (2.73) | -1.42 (2.47)

8. Secondary Outcome: Change in Body Mass Index
Description: Change from baseline (week 0) in body mass index (BMI). BMI was calculated based on body weight and height based on the formulae: BMI kg/m^2 = body weight (kg)/(Height (m) x Height (m)). Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Kilogram per square meter (kg/m^2)
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26 | -0.1 (0.7) | -0.4 (0.7) | -0.9 (1.1) | 0.0 (0.6) | -0.4 (0.6)
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52 | 0.0 (0.9) | -0.3 (0.8) | -1.1 (1.5) | 0.2 (0.7) | -0.4 (0.6)

9. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) in waist circumference. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Centimeters (cm)
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26 | 0.5 (3.9) | -0.6 (2.8) | -1.3 (3.8) | 0.0 (2.7) | -0.5 (2.1)
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52 | 0.2 (4.5) | -1.0 (2.8) | -2.7 (4.8) | 1.0 (3.7) | -0.9 (3.0)

10. Secondary Outcome: Change in Total Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in total cholesterol (measured as mmol/L) is presented as ratio to baseline. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Ratio of total cholesterol
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26 | 0.92 (9.6) | 0.93 (14.7) | 0.89 (12.6) | 0.94 (9.6) | 1.00 (12.3)
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52 | 0.99 (8.8) | 0.95 (10.6) | 0.93 (13.9) | 0.95 (9.0) | 1.01 (15.0)

11. Secondary Outcome: Change in HDL Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in high density lipoprotein (HDL) cholesterol (measured as mmol/L) is presented as ratio to baseline. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Ratio of HDL cholesterol
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26 | 0.97 (13.8) | 0.98 (14.7) | 0.96 (10.0) | 0.99 (11.5) | 1.03 (11.7)
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52 | 1.05 (12.2) | 1.01 (14.2) | 0.99 (12.2) | 0.98 (11.0) | 1.04 (10.5)

12. Secondary Outcome: Change in LDL Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in low density lipoprotein (LDL) cholesterol (measured as mmol/L) is presented as ratio to baseline. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Ratio of LDL cholesterol
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26 | 0.87 (14.6) | 0.89 (22.7) | 0.85 (18.2) | 0.91 (13.4) | 1.03 (19.8)
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52 | 0.99 (13.1) | 0.96 (15.5) | 0.91 (20.4) | 0.95 (12.3) | 1.06 (23.0)

13. Secondary Outcome: Change in VLDL Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in very low density lipoprotein (VLDL) cholesterol (measured as mmol/L) is presented as ratio to baseline. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Ratio of VLDL cholesterol
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26 | 1.02 (37.7) | 0.94 (37.2) | 0.93 (36.4) | 0.99 (33.1) | 0.87 (42.4)
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52 | 0.86 (32.3) | 0.84 (33.3) | 0.86 (45.3) | 0.87 (35.0) | 0.81 (45.6)

14. Secondary Outcome: Change in Triglycerides (Ratio to Baseline)
Description: Change from baseline (week 0) in triglycerides (measured as mmol/L) is presented as ratio to baseline. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Ratio of triglycerides
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26 | 1.03 (40.2) | 0.94 (38.3) | 0.93 (36.5) | 0.99 (33.5) | 0.87 (41.7)
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52 | 0.86 (32.3) | 0.84 (33.3) | 0.86 (45.4) | 0.87 (35.5) | 0.82 (44.7)

15. Secondary Outcome: Change in Fasting Insulin (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting insulin (measured as picomoles per liter [pmol/L]) is presented as ratio to baseline. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of insulin
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Ratio of insulin
  Week 26: number analyzed (Participants) | 43 | 45 | 42 | 45 | 41
  Week 26 | 1.19 (31.9) | 1.27 (49.0) | 1.10 (47.5) | 1.14 (37.1) | 0.92 (32.2)
  Week 52: number analyzed (Participants) | 38 | 43 | 40 | 41 | 34
  Week 52 | 1.07 (32.2) | 1.16 (38.5) | 1.04 (47.2) | 1.06 (35.9) | 0.93 (28.8)

16. Secondary Outcome: Change in Fasting C-peptide (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting C-peptide (measured as nanomoles per liter [nmol/L]) is presented as ratio to baseline. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of C-peptide
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Ratio of C-peptide
  Week 26: number analyzed (Participants) | 43 | 45 | 43 | 45 | 41
  Week 26 | 1.15 (23.2) | 1.24 (32.8) | 1.17 (35.0) | 1.18 (23.3) | 0.98 (20.7)
  Week 52: number analyzed (Participants) | 38 | 43 | 40 | 41 | 34
  Week 52 | 1.12 (24.9) | 1.19 (21.9) | 1.10 (34.2) | 1.11 (24.1) | 0.99 (20.6)

17. Secondary Outcome: Change in Fasting Glucagon (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting glucagon (measured as picograms per milliliter [pg/mL]) is presented as ratio to baseline. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of glucagon
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Ratio of glucagon
  Week 26: number analyzed (Participants) | 43 | 44 | 43 | 45 | 41
  Week 26 | 0.95 (16.3) | 0.89 (25.1) | 0.85 (22.9) | 0.91 (18.7) | 0.95 (16.0)
  Week 52: number analyzed (Participants) | 38 | 42 | 39 | 41 | 34
  Week 52 | 0.97 (14.7) | 0.95 (19.1) | 0.92 (19.8) | 0.93 (18.4) | 0.96 (14.2)

18. Secondary Outcome: Change in Fasting Pro-insulin (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting pro-insulin (measured as pmol/L) is presented as ratio to baseline. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of pro-insulin
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Ratio of pro-insulin
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26 | 0.69 (52.7) | 0.68 (56.1) | 0.51 (77.8) | 0.61 (49.0) | 0.85 (34.6)
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52 | 0.83 (46.6) | 0.78 (41.7) | 0.56 (68.6) | 0.72 (49.4) | 1.04 (37.9)

19. Secondary Outcome: Change in Fasting Pro-insulin/Insulin Ratio (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting pro-insulin/insulin ratio is presented as ratio to baseline. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of pro-insulin/insulin ratio
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Ratio of pro-insulin/insulin ratio
  Week 26: number analyzed (Participants) | 40 | 44 | 31 | 44 | 41
  Week 26 | 0.59 (42.7) | 0.54 (34.2) | 0.49 (42.4) | 0.55 (40.3) | 0.92 (29.1)
  Week 52: number analyzed (Participants) | 37 | 43 | 34 | 40 | 34
  Week 52 | 0.78 (39.1) | 0.67 (42.2) | 0.56 (39.6) | 0.69 (39.3) | 1.11 (29.2)

20. Secondary Outcome: Change in Insulin Resistance (HOMA-IR) (Ratio to Baseline)
Description: Change from baseline (week 0) in insulin resistance (measured as percentage of insulin resistance) by homeostatic model assessment index of insulin resistance (HOMA-IR) is presented as ratio to baseline. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of insulin resistance
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Ratio of insulin resistance
  Week 26: number analyzed (Participants) | 43 | 45 | 42 | 45 | 41
  Week 26 | 0.98 (44.7) | 1.02 (66.0) | 0.83 (58.5) | 0.86 (46.3) | 0.88 (43.8)
  Week 52: number analyzed (Participants) | 38 | 43 | 40 | 41 | 34
  Week 52 | 0.93 (44.9) | 0.95 (42.9) | 0.78 (62.0) | 0.82 (51.2) | 0.97 (38.6)

21. Secondary Outcome: Change in Beta-cell Function (HOMA-B) (Ratio to Baseline)
Description: Change from baseline (week 0) in beta-cell function (measured as percentage of beta-cell function) by homeostatic model assessment index of beta-cell function is presented as ratio to baseline. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26 and week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of beta-cell function
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Ratio of beta-cell function
  Week 26: number analyzed (Participants) | 43 | 45 | 42 | 45 | 41
  Week 26 | 1.71 (38.6) | 1.93 (41.2) | 1.95 (42.7) | 1.89 (40.2) | 1.00 (32.7)
  Week 52: number analyzed (Participants) | 38 | 43 | 40 | 41 | 34
  Week 52 | 1.36 (40.6) | 1.75 (47.2) | 1.86 (35.3) | 1.69 (42.2) | 0.89 (29.2)

22. Secondary Outcome: Participants Who Achieved HbA1c < 7.0% (53 mmol/Mol) ADA Target (Yes/no)
Description: Participants who achieved HbA1c <7.0% (53 millimoles per mole [mmol/mol]) according to American Diabetes Association (ADA) target, at week 26 and week 52. Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 26 and week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Participants
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26: Yes | 24 | 33 | 35 | 24 | 6
  Week 26: No | 19 | 12 | 9 | 21 | 35
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52: Yes | 19 | 29 | 33 | 20 | 4
  Week 52: No | 19 | 14 | 8 | 21 | 30

23. Secondary Outcome: Participants Who Achieved HbA1c Below or Equal to 6.5% (48 mmol/Mol), AACE Target (Yes/No)
Description: Participants who achieved HbA1c below or equal to 6.5% (48 mmol/mol), American Association of Clinical Endocrinologists target (Yes/No). Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 26 and week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Participants
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26: Yes | 13 | 24 | 28 | 16 | 2
  Week 26: No | 30 | 21 | 16 | 29 | 39
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52: Yes | 11 | 20 | 24 | 11 | 1
  Week 52: No | 27 | 23 | 17 | 30 | 33

24. Secondary Outcome: Participants Who Achieved HbA1c Below 7.0% (53 mmol/Mol) Without Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemia Episodes and no Weight Gain (Yes/No)
Description: Severe or BG-confirmed symptomatic hypoglycaemia is an episode that is severe according to the American Diabetes Association classification or blood glucose-confirmed by a plasma glucose value <3.1 mmol/L (56 milligrams per deciliter [mg/dL]) with symptoms consistent with hypoglycaemia. Number of participants who achieved HbA1c below 7.0% (53 mmol/mol) without severe or blood glucose confirmed symptomatic hypoglycaemia episodes and no weight gain (Yes/No). Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 26 and week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Participants
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26: Yes | 15 | 26 | 30 | 15 | 4
  Week 26: No | 28 | 19 | 14 | 30 | 37
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52: Yes | 12 | 24 | 28 | 9 | 4
  Week 52: No | 26 | 19 | 13 | 32 | 30

25. Secondary Outcome: Participants Who Achieved HbA1c Reduction Above or Equal to 1% (10.9 mmol/Mol) and Weight Loss Above or Equal to 3%
Description: Participants who achieved above or equal to 1% (10.9 mmol/mol) reduction in HbA1c and losing 3% or more of baseline body weight (Yes/No). Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 26 and week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Participants
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26: Yes | 7 | 11 | 21 | 5 | 3
  Week 26: No | 36 | 34 | 23 | 40 | 38
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52: Yes | 8 | 7 | 20 | 2 | 1
  Week 52: No | 30 | 36 | 21 | 39 | 33

26. Secondary Outcome: Participants Who Achieved Weight Loss Above or Equal to 5% (Yes/No)
Description: Participants losing 5% or more of baseline body weight (Yes/No). Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 26 and week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Participants
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26: Yes | 1 | 5 | 16 | 0 | 3
  Week 26: No | 42 | 40 | 28 | 45 | 38
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52: Yes | 1 | 5 | 17 | 2 | 2
  Week 52: No | 37 | 38 | 24 | 39 | 32

27. Secondary Outcome: Participants Who Achieved Weight Loss Above or Equal to 10% (Yes/No)
Description: Participants losing 10% or more of baseline body weight (Yes/No). Data based on on-treatment without rescue medication observation period is presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 26 and week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Participants
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26: Yes | 0 | 0 | 3 | 0 | 0
  Week 26: No | 43 | 45 | 41 | 45 | 41
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52: Yes | 0 | 1 | 6 | 0 | 0
  Week 52: No | 38 | 42 | 35 | 41 | 34

28. Secondary Outcome: Time to Additional Anti-diabetic Medication
Description: Presented results are the number of participants who had taken additional anti-diabetic medication anytime from week 0 to week 52. 'Additional anti-diabetic medication': use of new anti-diabetic medication for more than 21 days with the initiation at or after randomisation and before (planned) end-of-treatment. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Weeks 0 - 52
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Participants
  Up to Week 26 | 3 | 3 | 1 | 0 | 7
  Up to Week 52 | 8 | 6 | 4 | 4 | 15
Statistical Analysis 1: Comparison: Oral Semaglutide 3 mg vs Placebo; Time to initiation of additional anti-diabetic medication was analysed using a Cox proportional hazards model with treatment and stratification factor as categorical fixed effects and baseline HbA1c as covariate. Withdrawal for any reason or lost to follow-up contributed to the analysis as events (initiation of additional anti-diabetic medication). Censoring time was one day before planned end of treatment; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.2579, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.29 to 1.40] — Oral semaglutide 3 mg / Placebo
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Placebo; [analysis description as in outcome 28, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0052, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.25, 95% CI 2-sided [0.10 to 0.66] — Oral semaglutide 7 mg / Placebo
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 28, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0259, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.11 to 0.87] — Oral semaglutide 14 mg / Placebo
Statistical Analysis 4: Comparison: Oral Semaglutide 3 mg vs Liraglutide 0.9 mg; [analysis description as in outcome 28, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0674, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 2.70, 95% CI 2-sided [0.93 to 7.80] — Oral semaglutide 3 mg / Liraglutide 0.9 mg
Statistical Analysis 5: Comparison: Oral Semaglutide 7 mg vs Liraglutide 0.9 mg; [analysis description as in outcome 28, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.9087, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.32 to 3.54] — Oral semaglutide 7 mg / Liraglutide 0.9 mg
Statistical Analysis 6: Comparison: Oral Semaglutide 14 mg vs Liraglutide 0.9 mg; [analysis description as in outcome 28, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.6498, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.38 to 4.62] — Oral semaglutide 14 mg / Liraglutide 0.9 mg

29. Secondary Outcome: Time to Rescue Medication
Description: Presented results are the number of participants who had taken rescue medication anytime from week 0 to week 52. 'Rescue medication': use of new anti-diabetic medication as add-on to trial product and used for more than 21 days with the initiation at or after randomisation and before last day on trial product. Time to rescue medication was estimated based on data from on-treatment without rescue medication observation period.
Time Frame: Weeks 0 - 52
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Participants
  Up to Week 26 | 2 | 2 | 1 | 0 | 7
  Up to Week 52 | 7 | 5 | 4 | 3 | 15
Statistical Analysis 1: Comparison: Oral Semaglutide 3 mg vs Placebo; Time to initiation of rescue medication was analysed using a Cox proportional hazards model with treatment and stratification factor as categorical fixed effects and baseline HbA1c as covariate. Censoring time was one day before last day on trial product; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0219, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.14 to 0.86] — Oral semaglutide 3 mg / Placebo
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Placebo; [analysis description as in outcome 29, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0005, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.15, 95% CI 2-sided [0.05 to 0.44] — Oral semaglutide 7 mg / Placebo
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 29, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0098, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.23, 95% CI 2-sided [0.07 to 0.70] — Oral semaglutide 14 mg / Placebo
Statistical Analysis 4: Comparison: Oral Semaglutide 3 mg vs Liraglutide 0.9 mg; [analysis description as in outcome 29, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.1193, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 2.95, 95% CI 2-sided [0.76 to 11.46] — Oral Semaglutide 3 mg / Liraglutide 0.9 mg
Statistical Analysis 5: Comparison: Oral Semaglutide 7 mg vs Liraglutide 0.9 mg; [analysis description as in outcome 29, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.7147, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [0.31 to 5.56] — Oral Semaglutide 7 mg / Liraglutide 0.9 mg
Statistical Analysis 6: Comparison: Oral Semaglutide 14 mg vs Liraglutide 0.9 mg; [analysis description as in outcome 29, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.3765, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 1.97, 95% CI 2-sided [0.44 to 8.85] — Oral Semaglutide 14 mg / Liraglutide 0.9 mg

30. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event (AE) with onset in the on-treatment observation period (time period when a participant was on treatment with trial product, including the period after initiation of rescue medication, if any, and excluding any period after premature trial product discontinuation) assessed up to approximately 57 weeks (52 weeks treatment period + 5 weeks follow-up period).
Time Frame: Weeks 0 - 57
Population: Overall number of participants analyzed = safety analysis set (SAS) which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Adverse events
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Adverse events | 119 | 111 | 96 | 116 | 106

31. Secondary Outcome: Change in Amylase (Ratio to Baseine)
Description: Change in amylase (measured as units per liter [U/L]) is presented as ratio to baseline. Data based on on-treatment observation period is presented. The on-treatment observation period - time period when a participant was on treatment with trial product, including the period after initiation of rescue medication, if any and excluding any period after premature trial product discontinuation.
Time Frame: Week 0, week 26, week 52
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product. Number Analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Ratio of amylase
  Week 26: number analyzed (Participants) | 45 | 48 | 45 | 45 | 49
  Week 26 | 1.03 (20.1) | 1.10 (20.7) | 1.16 (30.9) | 1.07 (18.7) | 1.02 (18.9)
  Week 52: number analyzed (Participants) | 45 | 48 | 45 | 43 | 49
  Week 52 | 1.06 (18.9) | 1.10 (17.8) | 1.12 (18.0) | 1.06 (18.2) | 1.02 (16.7)

32. Secondary Outcome: Change in Lipase (Ratio to Baseine)
Description: Change in lipase (measured as U/L) is presented as ratio to baseline. Data based on on-treatment observation period is presented. The on-treatment observation period - time period when a participant was on treatment with trial product, including the period after initiation of rescue medication, if any and excluding any period after premature trial product discontinuation.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 31
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Ratio of lipase
  Week 26: number analyzed (Participants) | 45 | 48 | 45 | 45 | 49
  Week 26 | 1.25 (41.7) | 1.35 (34.5) | 1.61 (67.4) | 1.47 (52.1) | 1.04 (48.5)
  Week 52: number analyzed (Participants) | 45 | 48 | 45 | 43 | 49
  Week 52 | 1.29 (34.2) | 1.41 (45.8) | 1.47 (45.9) | 1.60 (46.8) | 1.03 (38.7)

33. Secondary Outcome: Change in Pulse Rate
Description: Change from baseline in pulse rate. Data based on on-treatment observation period is presented. The on-treatment observation period - time period when a participant was on treatment with trial product, including the period after initiation of rescue medication, if any and excluding any period after premature trial product discontinuation.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Beats per minute (beats/min)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Beats per minute (beats/min)
  Week 26: number analyzed (Participants) | 45 | 48 | 45 | 45 | 49
  Week 26 | 1 (7) | 2 (9) | 2 (8) | 2 (9) | 0 (8)
  Week 52: number analyzed (Participants) | 45 | 48 | 45 | 43 | 49
  Week 52 | 1 (7) | 3 (7) | 4 (10) | 2 (9) | 0 (7)

34. Secondary Outcome: Change in Blood Pressure
Description: Change from baseline in blood pressure (systolic [sBP] and diastolic [dBP]). Data based on on-treatment observation period is presented. The on-treatment observation period - time period when a participant was on treatment with trial product, including the period after initiation of rescue medication, if any and excluding any period after premature trial product discontinuation.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Millimeters of mercury (mmHg)
  Week 26: sBP: number analyzed (Participants) | 45 | 48 | 45 | 45 | 49
  Week 26: sBP | -3 (13) | -5 (12) | -2 (12) | -1 (13) | -4 (11)
  Week 52: sBP: number analyzed (Participants) | 45 | 48 | 45 | 43 | 49
  Week 52: sBP | -0 (12) | -1 (10) | -1 (10) | 1 (15) | -3 (9)
  Week 26: dBP: number analyzed (Participants) | 45 | 48 | 45 | 45 | 49
  Week 26: dBP | -0 (9) | -2 (7) | 1 (6) | -1 (9) | -3 (10)
  Week 52: dBP: number analyzed (Participants) | 45 | 48 | 45 | 43 | 49
  Week 52: dBP | -1 (8) | -0 (7) | -0 (7) | -0 (10) | -2 (8)

35. Secondary Outcome: Change in ECG Evaluation
Description: Electrocardiogram (ECG) was evaluated and interpreted by the investigator and categorised as normal, abnormal not clinically significant (NCS) or abnormal clinically significant (CS). The number of participants who had shifted from normal, abnormal NCS or abnormal CS ECG results from baseline (week 0) to week 26, week 52 is presented. Data based on in-trial observation period is presented. In-trial observation period - time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Participants
  Normal (week 0) to normal (week 26): number analyzed (Participants) | 38 | 41 | 39 | 40 | 41
  Normal (week 0) to normal (week 26) | 34 | 41 | 39 | 38 | 39
  Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 38 | 41 | 39 | 40 | 41
  Normal (week 0) to abnormal NCS (week 26) | 4 | 0 | 0 | 2 | 2
  Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 38 | 41 | 39 | 40 | 41
  Normal (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 0 | 0
  Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 6 | 6 | 7 | 5 | 7
  Abnormal NCS (week 0) to normal (week 26) | 3 | 1 | 3 | 1 | 1
  Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 6 | 6 | 7 | 5 | 7
  Abnormal NCS (week 0) to abnormal NCS (week 26) | 3 | 5 | 4 | 4 | 6
  Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 6 | 6 | 7 | 5 | 7
  Abnormal NCS (week 0) to abnormal CS (week 26) | 0 | 0 | 0 | 0 | 0
  Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 2 | 2 | 1 | 1 | 1
  Abnormal CS (week 0) to normal (week 26) | 2 | 0 | 0 | 0 | 0
  Abnormal CS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 2 | 2 | 1 | 1 | 1
  Abnormal CS (week 0) to abnormal NCS (week 26) | 0 | 0 | 0 | 0 | 1
  Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 2 | 2 | 1 | 1 | 1
  Abnormal CS (week 0) to abnormal CS (week 26) | 0 | 2 | 1 | 1 | 0
  Normal (week 0) to normal (week 52): number analyzed (Participants) | 38 | 41 | 39 | 39 | 41
  Normal (week 0) to normal (week 52) | 37 | 40 | 36 | 37 | 39
  Normal (week 0) to abnormal NCS (week 52): number analyzed (Participants) | 38 | 41 | 39 | 39 | 41
  Normal (week 0) to abnormal NCS (week 52) | 1 | 1 | 3 | 2 | 2
  Normal (week 0) to abnormal CS (week 52): number analyzed (Participants) | 38 | 41 | 39 | 39 | 41
  Normal (week 0) to abnormal CS (week 52) | 0 | 0 | 0 | 0 | 0
  Abnormal NCS (week 0) to normal (week 52): number analyzed (Participants) | 6 | 6 | 7 | 5 | 7
  Abnormal NCS (week 0) to normal (week 52) | 3 | 2 | 2 | 2 | 3
  Abnormal NCS (week 0) to abnormal NCS (week 52): number analyzed (Participants) | 6 | 6 | 7 | 5 | 7
  Abnormal NCS (week 0) to abnormal NCS (week 52) | 3 | 4 | 5 | 3 | 4
  Abnormal NCS (week 0) to abnormal CS (week 52): number analyzed (Participants) | 6 | 6 | 7 | 5 | 7
  Abnormal NCS (week 0) to abnormal CS (week 52) | 0 | 0 | 0 | 0 | 0
  Abnormal CS (week 0) to normal (week 52): number analyzed (Participants) | 2 | 2 | 1 | 1 | 1
  Abnormal CS (week 0) to normal (week 52) | 2 | 0 | 1 | 0 | 0
  Abnormal CS (week 0) to abnormal NCS (week 52): number analyzed (Participants) | 2 | 2 | 1 | 1 | 1
  Abnormal CS (week 0) to abnormal NCS (week 52) | 0 | 0 | 0 | 0 | 1
  Abnormal CS (week 0) to abnormal CS (week 52): number analyzed (Participants) | 2 | 2 | 1 | 1 | 1
  Abnormal CS (week 0) to abnormal CS (week 52) | 0 | 2 | 0 | 1 | 0

36. Secondary Outcome: Change in Physical Examination
Description: Physical examination included examination of cardiovascular system, nervous system (central and peripheral), gastrointestinal system including mouth, general appearence, head and neck (head, ears, eyes, nose, throat, neck), lymph node palpation, musculoskeletal system, respiratory system, skin and thyroid gland. Physical examination was performed by the investigator and categorised as normal, abnormal NCS or abnormal CS. Data based on in-trial observation period is presented. In-trial observation period - time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Baseline (Week -8), week 26, week 52
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Participants
  Week -8: Cardiovascular- Normal | 49 | 49 | 48 | 48 | 49
  Week -8: Cardiovascular- Abnormal NCS | 0 | 0 | 0 | 0 | 0
  Week -8: Cardiovascular- Abnormal CS | 0 | 0 | 0 | 0 | 0
  Week 26: Cardiovascular- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Cardiovascular- Normal | 46 | 49 | 47 | 45 | 49
  Week 26: Cardiovascular- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Cardiovascular- Abnormal NCS | 0 | 0 | 0 | 0 | 0
  Week 26: Cardiovascular- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Cardiovascular- Abnormal CS | 0 | 0 | 0 | 0 | 0
  Week 52: Cardiovascular- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Cardiovascular- Normal | 46 | 49 | 47 | 45 | 49
  Week 52: Cardiovascular- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Cardiovascular- Abnormal NCS | 0 | 0 | 0 | 0 | 0
  Week 52: Cardiovascular- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Cardiovascular- Abnormal CS | 0 | 0 | 0 | 0 | 0
  Week -8: Nervous system- Normal | 48 | 48 | 48 | 48 | 48
  Week -8: Nervous system- Abnormal NCS | 1 | 0 | 0 | 0 | 1
  Week -8: Nervous system- Abnormal CS | 0 | 1 | 0 | 0 | 0
  Week 26: Nervous system- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Nervous system- Normal | 45 | 48 | 47 | 45 | 48
  Week 26: Nervous system- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Nervous system- Abnormal NCS | 1 | 0 | 0 | 0 | 1
  Week 26: Nervous system- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Nervous system- Abnormal CS | 0 | 1 | 0 | 0 | 0
  Week 52: Nervous system- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Nervous system- Normal | 45 | 48 | 47 | 45 | 48
  Week 52: Nervous system- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Nervous system- Abnormal NCS | 1 | 0 | 0 | 0 | 1
  Week 52: Nervous system- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Nervous system- Abnormal CS | 0 | 1 | 0 | 0 | 0
  Week -8: Gastrointestinal sys- Normal | 46 | 47 | 47 | 47 | 48
  Week -8: Gastrointestinal sys- Abnormal NCS | 2 | 1 | 0 | 0 | 1
  Week -8: Gastrointestinal sys- Abnormal CS | 1 | 1 | 1 | 1 | 0
  Week 26: Gastrointestinal sys - Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Gastrointestinal sys - Normal | 44 | 47 | 45 | 44 | 48
  Week 26: Gastrointestinal sys- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Gastrointestinal sys- Abnormal NCS | 1 | 1 | 1 | 0 | 1
  Week 26: Gastrointestinal sys- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Gastrointestinal sys- Abnormal CS | 1 | 1 | 1 | 1 | 0
  Week 52: Gastrointestinal sys- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Gastrointestinal sys- Normal | 43 | 45 | 45 | 44 | 47
  Week 52: Gastrointestinal sys- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Gastrointestinal sys- Abnormal NCS | 2 | 3 | 1 | 0 | 2
  Week 52: Gastrointestinal sys- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Gastrointestinal sys- Abnormal CS | 1 | 1 | 1 | 1 | 0
  Week -8: General appearance- Normal | 47 | 47 | 47 | 47 | 46
  Week -8: General appearance- Abnormal NCS | 2 | 2 | 1 | 1 | 3
  Week -8: General appearance- Abnormal CS | 0 | 0 | 0 | 0 | 0
  Week 26: General appearance- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: General appearance- Normal | 44 | 47 | 45 | 44 | 46
  Week 26: General appearance- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: General appearance- Abnormal NCS | 2 | 2 | 2 | 1 | 3
  Week 26: General appearance- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: General appearance- Abnormal CS | 0 | 0 | 0 | 0 | 0
  Week 52: General appearance- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: General appearance- Normal | 43 | 48 | 46 | 44 | 46
  Week 52: General appearance- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: General appearance- Abnormal NCS | 2 | 1 | 1 | 1 | 3
  Week 52: General appearance- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: General appearance- Abnormal CS | 1 | 0 | 0 | 0 | 0
  Week -8: Head and neck- Normal | 44 | 45 | 44 | 45 | 46
  Week -8: Head and neck- Abnormal NCS | 5 | 1 | 1 | 3 | 3
  Week -8: Head and neck- Abnormal CS | 0 | 3 | 3 | 0 | 0
  Week 26: Head and neck- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Head and neck- Normal | 43 | 47 | 43 | 44 | 44
  Week 26: Head and neck- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Head and neck- Abnormal NCS | 3 | 0 | 1 | 1 | 3
  Week 26: Head and neck- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Head and neck- Abnormal CS | 0 | 2 | 3 | 0 | 2
  Week 52: Head and neck- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Head and neck- Normal | 42 | 47 | 43 | 44 | 44
  Week 52: Head and neck- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Head and neck- Abnormal NCS | 4 | 0 | 2 | 1 | 3
  Week 52: Head and neck- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Head and neck- Abnormal CS | 0 | 2 | 2 | 0 | 2
  Week -8: Lymph node- Normal | 49 | 49 | 48 | 48 | 49
  Week -8: Lymph node- Abnormal NCS | 0 | 0 | 0 | 0 | 0
  Week -8: Lymph node- Abnormal CS | 0 | 0 | 0 | 0 | 0
  Week 26: Lymph node- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Lymph node- Normal | 46 | 49 | 47 | 45 | 49
  Week 26: Lymph node- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Lymph node- Abnormal NCS | 0 | 0 | 0 | 0 | 0
  Week 26: Lymph node- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Lymph node- Abnormal CS | 0 | 0 | 0 | 0 | 0
  Week 52: Lymph node- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Lymph node- Normal | 46 | 49 | 47 | 45 | 49
  Week 52: Lymph node- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Lymph node- Abnormal NCS | 0 | 0 | 0 | 0 | 0
  Week 52: Lymph node- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Lymph node- Abnormal CS | 0 | 0 | 0 | 0 | 0
  Week -8: Musculoskeletal- Normal | 47 | 44 | 47 | 48 | 44
  Week -8: Musculoskeletal- Abnormal NCS | 2 | 3 | 0 | 0 | 4
  Week -8: Musculoskeletal- Abnormal CS | 0 | 2 | 1 | 0 | 1
  Week 26: Musculoskeletal- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Musculoskeletal- Normal | 42 | 45 | 46 | 43 | 42
  Week 26: Musculoskeletal- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Musculoskeletal- Abnormal NCS | 4 | 2 | 0 | 1 | 6
  Week 26: Musculoskeletal- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Musculoskeletal- Abnormal CS | 0 | 2 | 1 | 1 | 1
  Week 52: Musculoskeletal- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Musculoskeletal- Normal | 41 | 45 | 46 | 45 | 43
  Week 52: Musculoskeletal- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Musculoskeletal- Abnormal NCS | 5 | 2 | 0 | 0 | 6
  Week 52: Musculoskeletal- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Musculoskeletal- Abnormal CS | 0 | 2 | 1 | 0 | 0
  Week -8: Respiratory sys- Normal | 49 | 49 | 46 | 47 | 49
  Week -8: Respiratory sys- Abnormal NCS | 0 | 0 | 0 | 1 | 0
  Week -8: Respiratory sys- Abnormal CS | 0 | 0 | 2 | 0 | 0
  Week 26: Respiratory sys- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Respiratory sys- Normal | 46 | 48 | 45 | 44 | 49
  Week 26: Respiratory sys- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Respiratory sys- Abnormal NCS | 0 | 1 | 0 | 1 | 0
  Week 26: Respiratory sys- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Respiratory sys- Abnormal CS | 0 | 0 | 2 | 0 | 0
  Week 52: Respiratory sys- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Respiratory sys- Normal | 46 | 49 | 45 | 44 | 49
  Week 52: Respiratory sys- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Respiratory sys- Abnormal NCS | 0 | 0 | 0 | 1 | 0
  Week 52: Respiratory sys- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Respiratory sys- Abnormal CS | 0 | 0 | 2 | 0 | 0
  Week -8: Skin- Normal | 46 | 48 | 45 | 47 | 45
  Week -8: Skin- Abnormal NCS | 2 | 1 | 0 | 1 | 2
  Week -8: Skin- Abnormal CS | 1 | 0 | 3 | 0 | 2
  Week 26: Skin- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Skin- Normal | 44 | 47 | 44 | 43 | 45
  Week 26: Skin- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Skin- Abnormal NCS | 1 | 1 | 0 | 1 | 2
  Week 26: Skin- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Skin- Abnormal CS | 1 | 1 | 3 | 1 | 2
  Week 52: Skin- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Skin- Normal | 44 | 47 | 44 | 45 | 46
  Week 52: Skin- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Skin- Abnormal NCS | 1 | 1 | 0 | 0 | 2
  Week 52: Skin- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Skin- Abnormal CS | 1 | 1 | 3 | 0 | 1
  Week -8: Thyroid - Normal | 48 | 48 | 48 | 48 | 49
  Week -8: Thyroid- Abnormal NCS | 1 | 0 | 0 | 0 | 0
  Week -8: Thyroid- Abnormal CS | 0 | 1 | 0 | 0 | 0
  Week 26: Thyroid- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Thyroid- Normal | 45 | 48 | 47 | 45 | 49
  Week 26: Thyroid- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Thyroid- Abnormal NCS | 1 | 0 | 0 | 0 | 0
  Week 26: Thyroid- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 26: Thyroid- Abnormal CS | 0 | 1 | 0 | 0 | 0
  Week 52: Thyroid- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Thyroid- Normal | 45 | 48 | 47 | 45 | 49
  Week 52: Thyroid- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Thyroid- Abnormal NCS | 1 | 0 | 0 | 0 | 0
  Week 52: Thyroid- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Thyroid- Abnormal CS | 0 | 1 | 0 | 0 | 0

37. Secondary Outcome: Change in Eye Examination Category
Description: Eye examination was performed by the investigator and categorised as normal, abnormal not clinically significant (NCS) or abnormal clinically significant (CS). Data based on in-trial observation period is presented. In-trial observation period - time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week -8, Week 52
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Participants
  Week -8: Left eye- Normal | 39 | 45 | 37 | 37 | 39
  Week -8: Left eye- Abnormal NCS | 4 | 2 | 4 | 6 | 5
  Week -8: Left eye- Abnormal CS | 6 | 2 | 7 | 5 | 5
  Week 52: Left eye- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Left eye- Normal | 36 | 46 | 38 | 37 | 41
  Week 52: Left eye- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Left eye- Abnormal NCS | 4 | 2 | 5 | 5 | 3
  Week 52: Left eye- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Left eye- Abnormal CS | 6 | 1 | 4 | 3 | 5
  Week -8: Right eye- Normal | 42 | 46 | 36 | 38 | 39
  Week -8: Right eye- Abnormal NCS | 2 | 2 | 5 | 7 | 4
  Week -8: Right eye- Abnormal CS | 5 | 1 | 7 | 3 | 6
  Week 52: Right eye- Normal: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Right eye- Normal | 39 | 44 | 36 | 39 | 44
  Week 52: Right eye- Abnormal NCS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Right eye- Abnormal NCS | 2 | 2 | 7 | 5 | 3
  Week 52: Right eye- Abnormal CS: number analyzed (Participants) | 46 | 49 | 47 | 45 | 49
  Week 52: Right eye- Abnormal CS | 5 | 3 | 4 | 1 | 2

38. Secondary Outcome: Anti-semaglutide Binding Antibodies (Yes/no)
Description: Number of participants with the presence or absence (yes/no) of anti-semaglutide binding antibodies in blood anytime post-baseline (week 0) and up to week 57. This endpoint is applicable only to the reporting groups "Oral semaglutide 3 mg, Oral semaglutide 7 mg and Oral semaglutide 14 mg". Data based on the in-trial observation period was presented. The in-trial observation period - time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0 - 57
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 49 | 49 | 48
Participants
  Yes | 0 | 1 | 1
  No | 49 | 48 | 47

39. Secondary Outcome: Anti-semaglutide Neutralising Antibodies (Yes/no)
Description: Number of participants with the presence or absence (yes/no) of anti-semaglutide neutralising antibodies in blood anytime post-baseline (week 0) and up to week 57. This endpoint is applicable only to the reporting groups "Oral semaglutide 3 mg, Oral semaglutide 7 mg and Oral semaglutide 14 mg". Data based on the in-trial observation period is presented. The in-trial observation period - time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0 - 57
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 49 | 49 | 48
Participants
  Yes | 0 | 0 | 0
  No | 49 | 49 | 48

40. Secondary Outcome: Anti-semaglutide Binding Antibodies Cross Reacting With Native GLP-1 (Yes/no)
Description: Number of participants with the presence or absence (yes/no) of anti-semaglutide binding antibodies cross reacting with native GLP-1 in blood anytime post-baseline (week 0) and up to week 57. This endpoint is applicable only to the reporting groups "Oral semaglutide 3 mg, Oral semaglutide 7 mg and Oral semaglutide 14 mg". Data based on the in-trial observation period was presented. The in-trial observation period - time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0 - 57
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 49 | 49 | 48
Participants
  Yes | 0 | 0 | 1
  No | 49 | 49 | 47

41. Secondary Outcome: Anti-semaglutide Neutralising Antibodies Cross Reacting With Native GLP-1 (Yes/no)
Description: Number of participants with the presence or absence (yes/no) of anti-semaglutide neutralising antibodies cross reacting with native GLP-1 in blood anytime post-baseline (week 0) and up to week 57. This endpoint is applicable only to the reporting groups "Oral semaglutide 3 mg, Oral semaglutide 7 mg and Oral semaglutide 14 mg". Data based on the in-trial observation period was presented. The in-trial observation period - time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Week 0 - 57
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 49 | 49 | 48
Participants
  Yes | 0 | 0 | 0
  No | 49 | 49 | 48

42. Secondary Outcome: Anti-semaglutide Binding Antibody Levels
Description: This outcome measure is only applicable for the oral semaglutide treatment arms (3 mg, 7 mg and 14 mg). It is based on the data from participants who were measured with anti-semaglutide antibodies anytime during post-baseline visits (weeks 0-57). Results are presented as percentage of bound radioactivity-labelled semaglutide /total added radioactivity-labelled semaglutide (%B/T). Results are based on the data from the in-trial observation period. The in-trial observation period - time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication or premature discontinuation of trial product.
Time Frame: Weeks 0-57
Population: "Overall number of participants analyzed"=number of participants who were found positive for anti-semaglutide antibodies.
Measure: Mean (Standard Deviation); unit: %B/T
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 0 | 1 | 1
%B/T
  Week 4: number analyzed (Participants) | 0 | 0 | 0
  Week 8: number analyzed (Participants) | 0 | 1 | 0
  Week 8 |  | 1.58 (0.00) |
  Week 14: number analyzed (Participants) | 0 | 0 | 0
  Week 26: number analyzed (Participants) | 0 | 0 | 0
  Week 38: number analyzed (Participants) | 0 | 0 | 1
  Week 38 |  |  | 2.40 (0.00)
  Week 52: number analyzed (Participants) | 0 | 0 | 0
  Week 57: number analyzed (Participants) | 0 | 0 | 0

43. Secondary Outcome: Number of Treatment-emergent Severe or Blood Glucose-confirmed Symptomatic Hypoglycaemic Episodes
Description: Hypoglycaemic episodes defined as treatment-emergent if the onset of the episode occurs within the on-treatment observation period. Severe or BG-confirmed symptomatic hypoglycaemia is an episode that is severe according to the American Diabetes Association classification or blood glucose-confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Data based on on-treatment observation period was presented. The on-treatment observation period - time period when a participant was on treatment with trial product, including the period after initiation of rescue medication, if any and excluding any period after premature trial product discontinuation.
Time Frame: Week 0 - 57
Population: as for outcome 38
Measure: Number; unit: Episodes
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Episodes | 0 | 0 | 0 | 2 | 0

44. Secondary Outcome: Participants With Treatment-emergent Severe or Blood Glucose-confirmed Symptomatic Hypoglycaemic Episodes
Description: Number of participants with treatment emergent severe or blood glucose-confirmed symptomatic hypoglycaemic episodes. Hypoglycaemic episodes defined as treatment-emergent if the onset of the episode occurs within the on-treatment observation period. Severe or BG-confirmed symptomatic hypoglycaemia is an episode that is severe according to the American Diabetes Association classification or blood glucose-confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. Data based on on-treatment observation period was presented. The on-treatment observation period - time period when a participant was on treatment with trial product, including the period after initiation of rescue medication, if any and excluding any period after premature trial product discontinuation.
Time Frame: Weeks 0 - 57
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Participants | 0 | 0 | 0 | 2 | 0

45. Secondary Outcome: Semaglutide Plasma Concentration
Description: Semaglutide plasma concentration is presented. Samples for pharmacokinetic (PK) analysis were drawn at any time during the visit except for the visit at week 26 where samples were taken both pre-dose and 60-90 minutes post dosing. This endpoint is applicable only to the reporting groups, "Oral semaglutide 3 mg, Oral semaglutide 7 mg and Oral semaglutide 14 mg". Data based on on-treatment observation period was presented. The on-treatment observation period - time period when a participant was on treatment with trial product, including the period after initiation of rescue medication, if any and excluding any period after premature trial product discontinuation.
Time Frame: Week 26 and week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles per liter (nmol/L)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 45 | 48 | 45
Nanomoles per liter (nmol/L)
  Week 26 pre-dose | 3.7 (96.7) | 9.5 (80.1) | 20.6 (92.5)
  Week 26 post-dose | 5.3 (92.9) | 13.9 (86.3) | 30.7 (80.9)
  Week 52 | 3.2 (89.1) | 9.2 (96.9) | 20.0 (148.9)

46. Secondary Outcome: Change in SF-36: Sub-domains
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ questionnaire measured the HRQoL on 8 domains on individual scale ranges. The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. Change from baseline in the sub-domain scores is presented. A positive change score indicates an improvement since baseline. Data based on on-treatment without rescue medication observation period is presented.
Time Frame: Week 0, week 26, week 52
Population: Overall number of participants analyzed = FAS which comprised all randomised participants. Number Analyzed = number of participants with available data. On-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Score on a scale
  Week 26: Physical Functioning: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26: Physical Functioning | -0.22 (2.53) | -0.09 (1.93) | 0.04 (2.71) | 0.09 (2.01) | -0.14 (2.63)
  Week 52: Physical Functioning: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52: Physical Functioning | -0.31 (3.63) | 0.30 (2.37) | -0.00 (3.42) | -0.09 (2.11) | -0.00 (2.96)
  Week 26: Role-Physical: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26: Role-Physical | -1.79 (4.91) | 0.00 (3.48) | 0.05 (3.31) | 0.10 (3.51) | -0.86 (5.70)
  Week 52: Role-Physical: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52: Role-Physical | -2.14 (5.94) | 0.15 (4.84) | -0.86 (4.69) | -0.59 (3.55) | -0.58 (3.99)
  Week 26: Bodily Pain: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26: Bodily Pain | -2.02 (8.92) | -0.89 (5.93) | 1.18 (6.21) | 0.48 (7.09) | -0.19 (6.19)
  Week 52: Bodily Pain: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52: Bodily Pain | -2.43 (9.02) | -0.16 (7.78) | 0.03 (8.30) | 0.98 (7.09) | -0.79 (8.10)
  Week 26: General Health: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26: General Health | -2.43 (4.49) | 0.52 (4.29) | 0.41 (4.33) | -0.00 (5.87) | -0.08 (6.06)
  Week 52: General Health: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52: General Health | -0.99 (5.07) | -1.24 (5.38) | -0.47 (4.00) | 0.62 (6.34) | -0.99 (6.96)
  Week 26: Vitality: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26: Vitality | -2.85 (5.85) | -0.48 (4.83) | -1.49 (4.93) | -0.18 (6.07) | -1.99 (9.66)
  Week 52: Vitality: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52: Vitality | -1.93 (6.84) | -0.82 (6.63) | -1.06 (6.08) | -0.13 (6.17) | -1.60 (7.55)
  Week 26: Social Functioning: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26: Social Functioning | -0.11 (4.25) | 0.77 (3.94) | -0.45 (5.62) | -0.66 (5.12) | -1.20 (6.52)
  Week 52: Social Functioning: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52: Social Functioning | -0.78 (4.67) | -0.58 (3.92) | 0.00 (5.30) | -0.48 (4.53) | -1.16 (5.72)
  Week 26: Role-Emotional: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26: Role-Emotional | -1.60 (8.21) | -0.00 (6.03) | 0.35 (5.39) | -0.09 (5.72) | -1.12 (5.80)
  Week 52: Role-Emotional: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52: Role-Emotional | -0.70 (5.94) | 0.18 (2.63) | -0.47 (5.86) | -0.19 (4.67) | -1.80 (8.31)
  Week 26: Mental Health: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26: Mental Health | -1.90 (9.00) | 0.77 (5.56) | -2.36 (6.23) | 1.71 (6.70) | -2.17 (6.81)
  Week 52: Mental Health: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52: Mental Health | -2.41 (7.63) | -0.52 (7.38) | -1.69 (5.12) | 0.72 (5.82) | -1.31 (6.49)

47. Secondary Outcome: Change in SF-36: Physical Component Summary (PCS)
Description: Change in short form 36 v2.0 acute domain PCS from baseline (week 0) to week 56. SF-36v2™ questionnaire measured the HRQoL on 8 domains on individual scale ranges. It consists of 2 component summary measures that further summarize 8 health domain scales. The PCS measure is derived from domain scales of physical functioning, role-physical, bodily pain, and general health. The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. A positive change score indicates an improvement since baseline. Data based on on-treatment without rescue medication observation period is presented.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Score on a scale
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26 | -1.33 (4.56) | -0.38 (3.28) | 0.93 (3.49) | -0.14 (3.21) | 0.20 (4.11)
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52 | -1.28 (6.03) | -0.12 (4.30) | 0.02 (4.05) | 0.10 (3.42) | -0.10 (4.03)

48. Secondary Outcome: Change in SF-36: Mental Component Summary (MCS)
Description: Change in short form 36 v2.0 acute domain MCS from baseline (week 0) to week 56. SF- 36v2™ questionnaire measured the HRQoL on 8 domains on individual scale ranges. The MCS measure is derived from domain scales of vitality, social functioning, role emotional and mental health. The scores 0-100 (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. A norm-based score of 50 corresponds to the mean score and 10 corresponds to the standard deviation of the 2009 U.S. general population. A positive change score indicates an improvement since baseline. Data based on on-treatment without rescue medication observation period is presented.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Score on a scale
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26 | -1.81 (7.23) | 0.56 (5.62) | -1.61 (4.14) | 0.49 (5.09) | -2.18 (7.42)
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52 | -1.56 (6.63) | -0.58 (5.02) | -1.16 (4.80) | 0.10 (4.44) | -1.94 (7.43)

49. Secondary Outcome: Change From Baseline in DTR-QOL: Total Score
Description: Diabetes Therapy-Related QOL (DTR-QOL) questionnaire is a 29-item patient-reported survey of patient health that measures the influence of diabetes treatment on HRQoL on 4 domains on individual scale ranges: "Burden on social activities and daily activities", "Anxiety and dissatisfaction with treatment", "Hypoglycemia" and "Satisfaction with treatment" on a 7-point graded response scale. Higher item scores indicate a higher level of HRQoL for items 1-25. For items 26-29 a higher score indicates a lower level of HRQoL. The domain score is calculated from the mean score of the attribute items, and the scoring range is converted to 0 - 100. The total score, after simple addition of the item scores, is converted to 0 - 100 (best-case response = 100; worstcase response = 0). Data based on on-treatment without rescue medication observation period is presented.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Score on a scale
  Week 26: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26 | 6.67 (15.81) | 7.98 (11.47) | 11.22 (12.99) | 9.77 (14.46) | 4.18 (14.13)
  Week 52: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52 | 6.97 (14.47) | 5.52 (12.29) | 8.02 (14.09) | 7.12 (15.09) | 0.57 (16.53)

50. Secondary Outcome: Change From Baseline in DTR-QOL: Sub-domains
Description: DTR-QOL questionnaire is a 29-item patient-reported survey of patient health that measures the the influence of diabetes treatment on HRQoL. DTR-QOL questionnaire measured the HRQoL on 4 domains on individual scale ranges: "Burden on social activities and daily activities", "Anxiety and dissatisfaction with treatment", "Hypoglycemia" and "Satisfaction with treatment" on a 7-point graded response scale. Higher item scores indicate a higher level of HRQoL for items 1-25. For items 26-29 a higher score indicates a lower level of HRQoL. The domain score is calculated from the mean score of the attribute items, and the scoring range is converted to 0 - 100. W26 and W52 refer to week 26 and week 52 respectively. Data based on on-treatment without rescue medication observation period was presented. The on-treatment without rescue medication observation period - time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
Number analyzed (Participants) | 49 | 49 | 48 | 48 | 49
Score on a scale
  W26: Burden on social and daily activities: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  W26: Burden on social and daily activities | 5.75 (20.31) | 5.87 (13.06) | 7.90 (16.55) | 10.11 (17.38) | 6.91 (19.59)
  W52: Burden on social and daily activities: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  W52: Burden on social and daily activities | 9.31 (17.06) | 5.49 (15.19) | 3.94 (19.66) | 7.60 (18.73) | 2.90 (23.08)
  W26: Anxiety and dissatisfaction with treatment: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  W26: Anxiety and dissatisfaction with treatment | 6.49 (18.32) | 10.46 (15.27) | 14.68 (17.01) | 13.52 (20.99) | 1.83 (17.91)
  W52: Anxiety and dissatisfaction with treatment: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  W52: Anxiety and dissatisfaction with treatment | 4.93 (19.32) | 5.04 (16.52) | 10.52 (16.04) | 7.01 (20.45) | -2.94 (22.27)
  Week 26: Hypoglycemia: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26: Hypoglycemia | 8.33 (23.50) | 3.15 (18.08) | 9.19 (20.95) | 3.80 (26.53) | 7.42 (20.30)
  Week 52: Hypoglycemia: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52: Hypoglycemia | 5.81 (19.07) | 1.26 (18.51) | 8.13 (20.15) | 4.47 (22.94) | 6.00 (16.26)
  Week 26: Satisfaction with treatment: number analyzed (Participants) | 43 | 45 | 44 | 45 | 41
  Week 26: Satisfaction with treatment | 8.33 (16.39) | 14.72 (23.21) | 17.14 (25.10) | 7.13 (25.60) | -3.25 (24.96)
  Week 52: Satisfaction with treatment: number analyzed (Participants) | 38 | 43 | 41 | 41 | 34
  Week 52: Satisfaction with treatment | 4.61 (23.47) | 10.85 (24.74) | 16.16 (26.80) | 8.43 (22.64) | -5.39 (21.09)

ADVERSE EVENTS:
Time Frame: Week 0 to week 57 (52 weeks treatment period + 5 weeks follow-up period). Results are based on the safety analysis set (SAS), which comprised all randomised participants who received at least one dose of trial product.
Description: Serious adverse events and other AEs were based on the on-treatment observation period, i.e., the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. All-cause mortality were based on the in-trial observation period, i.e., the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Liraglutide 0.9 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49 | 0/48 | 0/48 | 0/49
Serious Adverse Events (participants affected / at risk) | 2/49 | 3/49 | 0/48 | 0/48 | 3/49
Other Adverse Events (participants affected / at risk) | 29/49 | 21/49 | 25/48 | 23/48 | 27/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 3 mg (N=49) | Oral Semaglutide 7 mg (N=49) | Oral Semaglutide 14 mg (N=48) | Liraglutide 0.9 mg (N=48) | Placebo (N=49)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 3 mg (N=49) | Oral Semaglutide 7 mg (N=49) | Oral Semaglutide 14 mg (N=48) | Liraglutide 0.9 mg (N=48) | Placebo (N=49)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5) | 6 (9) | 6 (6) | 9 (11) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (6) | 3 (5) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (2) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (8) | 1 (2) | 3 (3) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 10 (12) | 8 (12) | 9 (19) | 14 (21) | 14 (24)
Nausea (Gastrointestinal disorders) | 2 (2) | 5 (6) | 4 (4) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3) | 2 (3) | 2 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT03018028/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT03018028/SAP_001.pdf